CLINICAL TRIAL: NCT05126940
Title: Bedside Lung Ultrasonography by Emergency Department Nurses as an Aid for Identifying Heart Failure in Patients With Acute Dyspnea
Brief Title: Bedside Lung Ultrasonography by Nurses in Acute Dyspnea.
Acronym: LUS
Status: Completed | Type: Observational
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, professor, University of Monastir
Other Study IDs: LR12SP18
Record Dates: First submitted 2021-09-29; First posted 2021-11-19 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Dyspnea; Cardiac
Keywords: Lung ultrasound; heart failure; diagnosis; accuracy; nurses
MeSH Terms: conditions — Dyspnea; Heart Failure; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- nurses: ED nurses trained to perform LUS and blinded to the final diagnosis
  Interventions: Diagnostic Test: we perform a lung ultrasound to all the patients admitted for dyspnea independantly from the final diagnosis
- emergency physician: certified emergency physician who had accomplished a full mentoring program for "Ultra-Sound Life Support".
  Interventions: Diagnostic Test: we perform a lung ultrasound to all the patients admitted for dyspnea independantly from the final diagnosis

INTERVENTIONS:
Diagnostic Test: we perform a lung ultrasound to all the patients admitted for dyspnea independantly from the final diagnosis — Patients were placed in a semi-recumbent or supine position depending on their respiratory tolerance. For each side of the chest, 4 zones have to be assessed : 2 anterior and 2 lateral. The operator should calculate the number of B-lines when present .
  Other Names: lus

SUMMARY:
This study assesses the potential of lung ultrasonography to diagnose heart failure.

DETAILED DESCRIPTION:
Dyspnea is one of the most distressing situations for the patient . Emergency cases do not always present in conditions that are ideal for immediate diagnosis, which sometimes compromises outcome. Physical examination, laboratory findings and radiography are imperfect, resulting in a need for sophisticated test results that delay management.

Lung ultrasonography is becoming a standard tool in critical cases in the ED.

the investigators aim to perform ultrasonography on consecutive patients admitted to the ICU with dyspnea, comparing lung ultrasonography results on initial presentation with the final diagnosis by the nurses.

Three items were assessed: artifacts (horizontal A lines or vertical B lines indicating interstitial syndrome), lung sliding, and alveolar consolidation and/or pleural effusion, these items were grouped to assess ultrasound profiles.

the study aimed to evaluate the accuracy and reproducibility of B-lines testing assessed by emergency nurses after 12-h training in the diagnosis of HF in patients admitted to the emergency department with acute dyspnea.

ELIGIBILITY:
Inclusion Criteria:

* non traumatic dyspnea with the final diagnosis of heart failure

Exclusion Criteria:

* age less than 18 years
* impossibility to give consent to participate in the study
* post-traumatic dyspnea
* pregnant women
* need for endotracheal intubation or inotropic drugs
* patients who were deemed too unstable for sonography by the treating team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A convenience sampling approach, including all patients admitted to the ED for acute dyspnea as chief complaint, was used.
Sampling Method: Non-Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
the accuracy of LUS performed by nurses in the diagnosis of heart failure | 0 days
  the accuracy of LUS in the diagnosis of heart failure measured by sensitivity .
the Specificity of LUS by nurses in the diagnosis of heart failure | 0 days
  the accuracy of LUS in the diagnosis of heart failure measured by specificity.
the reproducibility of LUS in by nurses the diagnosis of heart failure | 0 days
  the accuracy of LUS in the diagnosis of heart failure measured by area under the roc curve
Agreement between nurses and expert's | 0 days
  Agreement between nurses and expert's interpretation was assessed by kappa agreement index for ordinal LUS scale classification

CONTACTS AND LOCATIONS:
Locations (1):
- Nouira Semir, Monastir, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided